CLINICAL TRIAL: NCT03045913
Title: Prospective Multicenter Observational Study for Evaluating Efficacy and Safety of GENOSS Sirolimus-eluting Stent in Patients With Coronary Artery Disease (GENOSS Registry)
Brief Title: Genoss DES Prospective Multicenter Registry
Status: Completed | Type: Observational
Sponsor: Young Jin Youn, MD, PhD (Other)
Collaborators: Genoss Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Young Jin Youn, MD, PhD, Professor, Yonsei University
Organization: Yonsei University (Other)
Other Study IDs: Yonsei University
Record Dates: First submitted 2017-01-23; First posted 2017-02-08 (Estimated); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia; Myocardial Infarction
Keywords: Observational registry; All-comers open label registry; Genoss DES; Multicenter; Stenting; Coronary Artery Disease; Coronary revascularization; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Genoss DES: Subject implanted Genoss DES for coronary artery disease
  Interventions: Device: Genoss DES

INTERVENTIONS:
Device: Genoss DES — The Genoss DES (Genoss, Korea) L-605 cobalt chromium (CoCr) platform with a strut thickness of 70 µm Sirolimus drug with concentration of 1.15µg/mm2 Abluminal biodegradable PLA and PLGA polymers.

SUMMARY:
This registry is a clinical post-market evaluation of the Genoss DES in subjects requiring coronary revascularization with Drug Eluting Stents (DES).

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) is the main stream of treatment of coronary artery disease. Drug-eluting stents (DES) have dramatically reduced the rates of restenosis and target lesion revascularization (TLR) compared with bare-metal stents (BMS). Newer-generation DES with a durable polymer such as Xience (Abbott, US) and Resolute (Medtronic, US) were widely used. However, the concern about late stent thrombosis due to hypersensitivity reaction from the polymer is still existed. Recently, DES with a biodegradable polymer such as Biomatrix (Biosensors, Switzerland), Nobori (Terumo, Japan), Orsiro (Biotronik, Switzerland), and Synergy (Boston Scientific, US) was rapidly adopted and it is expected to reduce the late stent thrombosis.

Recently, new biodegradable DES with thin struts was developed in South Korea. The Genoss DES (Genoss, Korea) has an L-605 cobalt chromium (CoCr) platform with a strut thickness of about 70 µm and the stent is coated a combination of Sirolimus drug with concentration of 1.15µg/mm2 and an abluminal biodegradable PLA and PLGA polymers.

This study is conducted to evaluate efficacy and safety of Genoss DES in the treatment of patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 19 years
* Subject implanted Genoss DES within 1 month
* Subject has signed informed consent for data release
* Subject is geographically stable and willing to participate at all follow-up assessments

Exclusion Criteria:

* Subject did not sign informed consent for data release
* Known intolerance to aspirin, clopidogrel, ticlopidine, heparin or any other anticoagulation / antiplatelet therapy required for PCI, cobalt chromium, Sirolimus or contrast media
* Pregnancy
* Subject with life expectancy less than 12 months
* Subject with cardiogenic shock
* Planned surgery within 12 months of PCI unless dual antiplatelet therapy will be maintained
* Currently participating in another study and primary endpoint is not reached yet.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-comers patient population with all subjects requiring coronary revascularization with a Drug Eluting Stent (DES)
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2016-11-18 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Device-oriented composite end point (TLF) | 12 months
  Composite of cardiac death, any myocardial infarction not clearly attributable to a nontarget vessel, and clinically indicated target-lesion revascularization

SECONDARY OUTCOMES:
Patient-oriented composite end point | 12 months
  Composite of any death, any myocardial infarction, and any revascularization
Cardiac death | 12 months
  Any death due to proximate cardiac cause, unwitnessed death and death of unknown cause, and all procedure-related deaths, including those related to concomitant treatment
Non-cardiac death | 12 months
  Any death not covered by the cardiac death
Any myocardial infarction | 12 months
  New symptom Symptoms suggestive of ischemia + increased cardiac enzyme (Troponin >URL or CKMB >URL) or New ST elevation or LBBB
Any myocardial infarction not clearly attributable to a nontarget vessel | 12 months
  Any myocardial infarction not clearly attributable to a nontarget vessel
Any revascularization | 12 months
  Any repeat revascularization including all target and nontarget vessel
Clinically indicated target-lesion revascularization | 12 months
  Any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. The target lesion is defined as the treated segment from 5 mm proximal to the stent and to 5 mm distal to the stent.
Clinically indicated target-vessel revascularization | 12 months
  any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion, which includes upstream and downstream branches and the target lesion itself.
ARC defined stent thrombosis | 12 months
  * Definite stent thrombosis
    * Angiographic confirmation of stent thrombosis
    * Pathological confirmation of stent thrombosis
  * Probable stent thrombosis
    - Clinical definition of probable stent thrombosis is considered to have occurred after intracoronary stenting in the following cases:
  * Possible stent thrombosis - Clinical definition of possible stent thrombosis is considered to have occurred with any unexplained death from 30 days after intracoronary stenting until end of trial follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Junghan Yoon, MD, PhD, Principal Investigator — Wonju Severance Christian Hospital
Locations (17):
- South Korea (17):
  - Chungbuk National University Hospital, Cheongju-si, Chungcheongbuk
  - Dankook University Hospital, Cheonan, Chungcheongnam
  - Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do
  - Kangwon National University Hospital, Chuncheon, Gangwon-do
  - Gangneung Asan Hospital, Gangneung, Gangwon-do
  - Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggi-do
  - Myongji Hospital, Hanyang University College of Medicine, Goyang-si, Gyeonggi-do
  - National Health Insurance Service Ilsan Hospital, Goyang-si, Gyeonggi-do
  - CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Kosin University Gospel Hospital, Busan
  - Gachon University Gil Medical Center, Incheon
  - Ewha Womans University Mokdong Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Kangnam Sacred Heart Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Severance Cardiovascular Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No